CLINICAL TRIAL: NCT00001306
Title: Autoimmune Premature Ovarian Failure: A Controlled Trial of Alternate-Day Prednisone Therapy
Brief Title: Steroid Therapy in Autoimmune Premature Ovarian Failure
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920223; 92-CH-0223
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-12-12

CONDITIONS: Autoimmune Disease; Infertility; Premature Ovarian Failure
Keywords: Infertility; Ovulation; Autoimmune; Follicle; Menopause; Biopsy; Glucocorticoids; Premature Ovarian Failure; Amenorrhea; Ovarian Failure; POF
MeSH Terms: conditions — Autoimmune Diseases; Infertility; Primary Ovarian Insufficiency; Amenorrhea

SUMMARY:
No therapy for infertile patients with premature ovarian failure has been proven effective. Some anecdotal reports have suggested that high dose, long term prednisone (steroid) therapy may be useful in treating autoimmune ovarian failure. However, prednisone, when used in high-doses for long periods of time has substantial side effects, including aseptic necrosis of bone where portions of bone die without the presence of infection and are surrounded by healthy tissue. Aseptic necrosis of bone often requires major surgical treatment. Even with this known level of risk, patients with premature ovarian failure are being treated based on this anecdotal evidence.

This study will test the hypothesis that a lower risk therapy (alternate-day, lower dose, shorter-term prednisone) will cause a remission of autoimmune ovarian failure. There is no reliable blood test to identify patients who have premature ovarian failure. Therefore, all patients must undergo a laparoscopic ovarian biopsy to confirm the presence of an auto immune reaction in the ovaries (autoimmune oophoritis). Laparoscopy is a surgical procedure that allows doctors to explore the abdomen using a camera-like device called a laparoscope. The procedure has been used clinically by some reproductive endocrinologists to identify patients with premature ovarian failure who have an autoimmune mechanism for the disorder.

The treatment will be deemed successful based on the return of ovulation as determined by weekly serum progesterone levels.

DETAILED DESCRIPTION:
Autoimmune oophoritis is a distinct clinical entity and a known cause of premature ovarian failure. It is characterized by the presence of circulating adrenal antibodies. No therapy for infertile patients with premature ovarian failure due to autoimmune oophoritis has been proven effective by prospective controlled study. Anecdotal reports have suggested that high-dose, long-term prednisone therapy may be useful in treating autoimmune ovarian failure. However, prednisone, when used in high-dose for a long-term has substantial side effects, including aseptic necrosis of bone requiring major surgical intervention. Despite this risk, patients with premature ovarian failure are being treated based on this anecdotal evidence. We are aware of two patients with premature ovarian failure who developed aseptic necrosis of bone on high-dose, long-term prednisone therapy administered elsewhere.

This protocol will test the hypothesis that a lower risk therapy (alternate-day, lower dose, shorter-term prednisone) will induce remission of ovarian failure caused by autoimmune oophoritis. The protocol will use a double-masked, placebo-controlled design. Patients with premature ovarian failure who have serologic evidence of steroidogenic cell autoimmunity will be candidates. Successful outcome will be defined as a return of ovulation as determined by weekly serum progesterone levels. The hypothesis that short-term, alternate-day prednisone therapy restores ovulation will be tested with an equality of proportions test comparing the proportion of patients who ovulate during placebo with the proportion of patients who ovulate during prednisone therapy.

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA:

Women 18 to 39 years of age with premature ovarian failure who meet the following requirements will be candidates for the study:

At least a four month history of amenorrhea not due to pregnancy,

Clearly elevated gonadotropins with a serum FSH greater than or equal to 40 IU/L on two separate occasions at least one month apart,

Positive adrenal or ovarian antibodies demonstrated by indirect immuno-fluorescence using monkey tissue as substrate or other laboratory evidence of steroidogenic cell autoimmunity such as the presence of antibodies against 21-hydroxylase,

No evidence for genetic, metabolic, toxic, or iatrogenic cause of the ovarian failure,

No medical contraindication to glycocorticoid therapy,

No glycocorticoid therapy taken in the past year (patients on appropriate replacement therapy for Addison's disease are not excluded),

No medical contraindication to pregnancy.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 1992-07-10; Study Completion 2011-12-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Maity R, Caspi RR, Nair S, Rizzo LV, Nelson LM. Murine postthymectomy autoimmune oophoritis develops in association with a persistent neonatal-like Th2 response. Clin Immunol Immunopathol. 1997 Jun;83(3):230-6. doi: 10.1006/clin.1997.4338. PMID 9175911
- [Background] Anasti JN, Flack MR, Froehlich J, Nelson LM. The use of human recombinant gonadotropin receptors to search for immunoglobulin G-mediated premature ovarian failure. J Clin Endocrinol Metab. 1995 Mar;80(3):824-8. doi: 10.1210/jcem.80.3.7883837.
- [Background] Kim TJ, Anasti JN, Flack MR, Kimzey LM, Defensor RA, Nelson LM. Routine endocrine screening for patients with karyotypically normal spontaneous premature ovarian failure. Obstet Gynecol. 1997 May;89(5 Pt 1):777-9. doi: 10.1016/s0029-7844(97)00077-x. PMID 9166320